CLINICAL TRIAL: NCT02896803
Title: A Phase II Trial of Bolus Fluorouracil and Oxaliplatin (mFLOX) as First-line Regimen for Patients With Unresectable or Metastatic Pancreatic Cancer Not Eligible for Infusional Fluorouracil, Irinotecan and Oxaliplatin
Brief Title: Fluorouracil and Oxaliplatin as First-line for Advanced Pancreatic Cancer
Acronym: PanFLOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 869/15
Record Dates: First submitted 2016-08-29; First posted 2016-09-12 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic Cancer; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): mFLOX
  Interventions: Drug: mFLOX

INTERVENTIONS:
Drug: mFLOX — 5-fluorouracil 500 mg/m2 and folinic acid 20 mg/m2 infused both bolus weekly for 6 weeks (d1, 8,15, 22, 29 and 36) and oxaliplatin 85 mg / m2 infused over 2 hours at weeks 1,3 and 5 (d1,15 and 29). The scheme will be repeated every 8 weeks.
  Other Names: 5-fluorouracil and oxaliplatin

SUMMARY:
Patients with locally advanced or metastatic pancreatic adenocarcinoma not eligible for infusional fluorouracil, irinotecan and oxaliplatin (FOLFIRINOX) (PPS 2 or hyperbilirubinemia, among other causes) will be treated with mFLOX regimen (fluorouracil bolus and oxaliplatin). The primary endpoint is to assess the objective response rate according to RECIST criteria (version 1.1) and the secondary endpoints are time until clinical or radiological progression, overall survival, toxicity profile.

DETAILED DESCRIPTION:
Currently, FOLFIRINOX is considered the standard treatment for PS 0 or 1 patients with advanced pancreatic carcinoma. However, due to excessive toxicity dose reductions and interruptions in the treatment toxicity are frequent. So, for those not eligible patients (PS 2 or 3, hyperbilirubinemia, among other causes), alternative schemes as gemcitabine alone are the standard approach .

This study aims to evaluate the efficacy and safety of the mFLOX regimen (fluorouracil bolus and oxaliplatin) as first-line regimen for advanced pancreatic adenocarcinoma not eligible for FOLFIRINOX.

The primary endpoint is to assess the objective response rate according to RECIST criteria (version 1.1) and the secondary endpoints are time until clinical or radiological progression, overall survival, toxicity profile.

It has been estimated an n=34 for a response rate of 20%, compared to the historical control of 7% with gemcitabine alone (Von Hoff et al.), with an alpha error of 5% and power of 80%. Considering a rate of 10% of dropout, our sample will be 37 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic adenocarcinoma, confirmed by biopsy and histological material available for review
* Unresectable primary tumor considered by the team assistant or metastatic disease
* Aged between 18 and 75 at the time of study entry
* Naïve patients of palliative chemotherapy, admitted for treatment at the Institute of the São Paulo State Cancer (ICESP)
* Patients with performance status 0 or 1, not candidates to receive chemotherapy with FOLFIRINOX or performance status 2.
* No significant organ dysfunction defined as: Hb> 9 g / dL, platelets> 100,000 / microliter (mcL), neutrophils> 1500 / mcL, clearance of creatinine (ClCr) > 50 ml / min, total bilirubin <5 mg/dl, serum alanine transaminase (ALT) and aspartate transaminase (AST) <2.5 x upper limit of normal (ULN) (or <5 x ULN if liver metastases present)
* Able to read and sign an informed consent form.

Exclusion Criteria:

* Use of prior chemotherapy with other agents, except adjuvant chemotherapy with gemcitabine monotherapy since completed more than 6 months
* Absence of histological material available to local review (eg diagnostic fine needle aspiration (FNA) or cytology)
* Previous use of radiotherapy in the primary tumor or a metastasis site that will serve as target lesion to assess response to treatment
* Diagnosis of malignancy other activity except non-melanoma skin cancer
* Clinical evidence of metastasis in the central nervous system active meningeal carcinomatosis or severe chronic disease patients (cirrhosis, heart failure New York Heart Association Functional Classification (NYHA) III or IV, chronic obstructive pulmonary disease (COPD) oxygen-dependent or chronic kidney disease requiring dialysis)
* Pregnant or breastfeeding
* Patients with HIV / AIDS story on anti-retroviral therapy
* Patients with peripheral neuropathy grade> 2 (CTCAE v4.03)
* Medium or large surgery in the last 4 weeks. For example, biliary derivation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2016-08; Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | Through the study, every 14-16 weeks, until an average of 6 months
  Response rate will be evaluated according RECIST criteria version 1.1

SECONDARY OUTCOMES:
Time to progression | Through the study, every 14-16 weeks, until an average of 6 months
  CT scans will be performed every 14-16 weeks, until disease progression (according to RECIST criteria version 1.1) or death, an average of 6 months.
Overall survival | Through the study, an average of 10 months
  It is defined as a time between entry in the trial and death
Toxicities according CTCAE v4.03 | Through the treatment, every visit, an average of 6 months
  Toxicities will be evaluated every visit, according CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Castria, MD PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No